CLINICAL TRIAL: NCT05287815
Title: Determination of Health Care Needs of Elderly Individuals According to the Omaha Classification System and Investigation of the Effects of Implemented Nursing Interventions on Healthy Lifestyle Behaviors and Quality of Life
Acronym: health elderly
Status: Recruiting | Type: Observational
Sponsor: Nazmiye Güney (Other)
Collaborators: Eastern Mediterranean University (Other)
Responsible Party: Sponsor-Investigator, Nazmiye Güney, msc, Eastern Mediterranean University
Organization: Eastern Mediterranean University (Other)
Other Study IDs: ETK00-2022-0187; gulten sucu dag (Other: eastern mediterrenean university)
Record Dates: First submitted 2022-02-27; First posted 2022-03-18 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Nurse-Patient Relations
Keywords: health, elderly,nurse
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: experimental(30 people) groups health education will be given by making a home visit
  Interventions: Behavioral: training/observation
- 2: control(30 people) no intervention
  Interventions: Behavioral: training/observation

INTERVENTIONS:
Behavioral: training/observation — In the study, elderly individuals who met the sampling criteria and accepted to participate in the study were 30 in the experimental group and 30 in the control group, using the stratified randomization method to control and balance the effects of age (65-75 years, 76 and over) and gender (female and male) variables. It will be planned to be an elderly individual. Computer-assisted randomization, which is one of the simple randomization methods, was assigned to the groups according to the determined.
  Other Names: omaha system

SUMMARY:
As in the whole world, there is an increase in the elderly population in the TRNC. However, no systematic care is provided for the registration and follow-up of elderly individuals. In this study, it is aimed to determine the health care needs of the elderly with a systematic method with the Omaha Classification System (OSS), which is used in the home care system in the world and in Turkey, and to examine the effectiveness of the nursing interventions applied according to the health care needs of the elderly people. With this method, it is thought that the continuity of monitoring and monitoring the health care needs of elderly individuals with a systematic approach will be ensured.

DETAILED DESCRIPTION:
As in the whole world, there is an increase in the elderly population in the TRNC. However, no systematic care is provided for the registration and follow-up of elderly individuals. In this study, it is aimed to determine the health care needs of the elderly with a systematic method with the Omaha Classification System (OSS), which is used in the home care system in the world and in Turkey, and to examine the effectiveness of the nursing interventions applied according to the health care needs of the elderly people. With this method, it is thought that the continuity of monitoring and monitoring the health care needs of elderly individuals with a systematic approach will be ensured.

Thus, it will be ensured that nursing interventions for the health care needs of elderly individuals are planned and implemented, and the nursing interventions applied for the field of health behaviors they live will be planned. In line with the data to be obtained as a result of the research, it is aimed to establish a system that will provide an opportunity to provide quality nursing care aimed at improving the health of the elderly, which is an important area of public health nurses in the TRNC.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old self care

Exclusion Criteria:

* comminication barrier mentally handicapped

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 65 years old male and female elderly people
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Omaha Classification System: Nursing Intervention Chart | may 2021-april 2022
  Omaha Classification System: Nursing Intervention Chart (HGŞ), Turkish adaptation was made by Erdoğan and Esin (14). HGŞ; list of nursing interventions. It is organized according to the individual problems that the nurse defines in the PSL. Care plans are drawn up in line with the intervention categories of this scheme. Intervention categories consist of four parts: health education, guidance and counseling, treatment and procedure, case management and surveillance(14).
  In the reliability analysis of the Omaha Nursing Classification System; The cronbach alpha value was evaluated by kappa analysis and the Kappa value of the Nursing Interventions Chart was determined as 0.78 (Erdogan, S., & Esin, NM (2006). The Turkish version of the Omaha System: Its use in practice-based family nursing education. Nurse Education Today , 26(5), 396-402).
  Omaha Classification System: Nursing Intervention Chart (HGŞ), Turkish adaptation was made by Erdoğan and Esin (2006) (Erdoğan and Esin, 2006). HGŞ;
Healthy Lifestyle Behaviors Scale II | may 2021-april 2022
  The HLBD scale measures the health-promoting validity and reliability of the Healthy Lifestyle Behaviors Scale II was performed by Bahar et al. (2008) and Pınar et al. (2009). In the study of Bahar et al., the cronbach alpha value of the scale was found to be .92, and in the study of Pınar et al., the cronbach alpha value of the scale and all its sub-dimensions was found above .70 (Pinar et al.2009).
  SYBD II scale consists of 52 items and six sub-dimensions. These; spiritual development, interpersonal relationships, nutrition, physical activity, health responsibility and stress management. The scale is a 4-point Likert-type scale that is evaluated in the categories never (1), sometimes (2), often (3), and regularly (4)

CONTACTS AND LOCATIONS:
Locations (1):
- Nazmiye, Famagusta, Mutluyaka, Cyprus

IPD SHARING:
Plan to Share IPD: No